CLINICAL TRIAL: NCT03842943
Title: Neoadjuvant Combination Immunotherapy for Stage III Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Michael Egger, Principal Investigator, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 181095
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination T-VEC/Pembrolizumab (Experimental): Pre-operative talimogene laherparepvec (T-VEC) with Pembrolizumab
  T-VEC - intra-lesional injection into palpable lymph nodes every 3 weeks for 6 months, or until complete response of target tumors.
  Pembrolizumab - administered intravenously every 3 weeks for 6 months, then every 3 weeks for one year in the adjuvant setting following complete lymph node dissection.
  Interventions: Drug: Pembrolizumab; Drug: Talimogene Laherparepvec

INTERVENTIONS:
Drug: Pembrolizumab — Preoperative infusions
  Other Names: Keytruda
Drug: Talimogene Laherparepvec — Preoperative intralesional injection
  Other Names: T-VEC; Imlygic

SUMMARY:
Determine safety and efficacy of pre-operative combination immunotherapy with Talimogene Laherparepvec (T-VEC)/Pembrolizumab given prior to complete lymph node dissection in resectable stage 3 cutaneous melanoma with clinically apparent lymph node metastases.

DETAILED DESCRIPTION:
This is a single arm Phase 2 study of pre-operative combination immunotherapy with pembrolizumab and T-VEC given for 6 months prior to complete lymph node dissection for stage 3 resectable cutaneous melanoma with clinically apparent lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, any race or sex, who have pathologically confirmed cutaneous melanoma
* ECOG performance status of 0 or 1
* Adequate hematologic, hepatic, renal and coagulation function
* Must have measurable disease and have an injectable target lymph node for intralesional therapy administration
* Primary melanoma has been resected
* Pathologically confirmed resectable stage III disease, clinically apparent. Resectability is at the discretion of the treating surgeon who is a melanoma specialist.
* Stage III disease can be at time of diagnosis of primary melanoma or a recurrence after initial treatment of stage I-II disease.
* BRAF mutant or wild type allowed (mutations status not necessary for enrollment)
* Signed, written informed consent

Exclusion Criteria:

* Cannot have metastatic (AJCC M1) disease
* No primary mucosal or uveal melanoma
* No evidence of melanoma associated with immunodeficiency state or history or other malignancies (other than non-melanoma skin cancer) within the past 3 years
* May not have been previously treated with T-VEC, any other oncolytic virus, pembrolizumab, or any other PD-1, PD-L1, or PD-L2 inhibitor
* Must not have a history or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, document history of autoimmune disease or syndrome requiring systemic treatment in the past two years (i.e. use of disease modifying agents, steroids, or immunosuppressive agents) except vitiligo or resolved childhood asthma/atopy, or evidence of clinically significant immunosuppression
* Must not have active herpetic skin lesions or prior complications of herpetic infection and must not require intermittent or chronic treatment with an anti-herpetic drug (e.g. acyclovir) other than intermittent topical use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 6 months
  Pathologic response rate in the regional nodal basin assessed after complete lymph node dissection

SECONDARY OUTCOMES:
Safety and Tolerability of Preoperative T-VEC/pembrolizumab: Adverse events and Serious Adverse Events | Every 3-6 weeks during the combination treatment period, and every 3 months after surgery through study completion, up to 5 years
  Adverse events and Serious Adverse Events will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Michael Egger, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided